CLINICAL TRIAL: NCT00289393
Title: Response Shift in Patient Expectations and Functional Outcome Following Posterior Lumbar Spinal Surgery for Degenerative Spinal Disorders
Brief Title: Response Shift in Patient Expectations and Functional Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: REB #151-2004
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Spinal Injuries
MeSH Terms: conditions — Spinal Injuries | interventions — Physicians

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Behavioral: Perceived outcome by both patient and physician

SUMMARY:
The purpose of this study is to evaluate the results of elective lumbar spinal surgery as it relates to shifting patient expectations for outcome. Patients undergoing elective posterior spinal surgery for degenerative conditions of the spine at SWCHSC will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of a degenerative condition of the lumbar spine undergoing posterior lumbar spinal surgery at Sunnybrook and Women's College Health Sciences Centre
* Patients who have had previous lumbar surgery

Exclusion Criteria:

* Traumatic or neoplastic surgical conditions of the lumbar spine

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Joel Finkelstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada